CLINICAL TRIAL: NCT06748235
Title: Effects of Comprehensive Hand Repetition Intensive Strength Training on Upper LIMB Function in Children With Cerebral Palsy
Brief Title: Comprehensive Hand Repetation Intensive Strength Training on Upper Limb in Children With Cerebral Palsy
Acronym: CHRIST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR/AHS/24/NISHA
Record Dates: First submitted 2024-11-03; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Cerebral Palsy (CP)
Keywords: Cerebral palsy; Muscle strength; Upper extremity
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: It will be randomized control trial in which non probability convenient sampling will be used. Two groups of 6-12 age will be formed in which participants will be randomly divided. Group A will be receive Group-Task-Oriented Training. Group B will be receive routine therapy
Who Masked: Participant
Masking Description: participant will get separate treatment protocol and possible efforts will be put to mask the both group about the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group will received Comprehensive Hand Repetitive Intensive Strength Training (Experimental): Physical Therapy 60 minutes per session, three sessions a week, at a total of 30 sessions per ten weeks. Comprehensive hand repetitive intensive strength training included treadmill training for the upper limb with body weight supporting the using upper limb. The posture of an arm swing was to maintain the joints of the elbows and wrist as much as possible, and the shoulder joint was allowed to be flexed by 160 degrees.
  Interventions: Other: Intensive Strength Training
- Routine Physical Therapy (Other): control will received 60 minutes per a session, three sessions a week, at a total of 30 sessions per 10 weeks by creating a home program, which consisted of a total of 8 exercises that enhanced the muscular strength of the upper limb including the triceps brachii and extensor carpi radialis, and conveyed an effect of reaching the muscles out.
  Interventions: Other: Routine Physical Therapy

INTERVENTIONS:
Other: Intensive Strength Training — Comprehensive Hand Repetitive Intensive Strength Training and Routine Physical Therapy 60 minutes per session, three sessions a week, at a total of 30 sessions per ten weeks. Comprehensive hand repetitive intensive strength training included treadmill training for the upper limb with body weight supporting the using upper limb. The posture of an arm swing was to maintain the joints of the elbows and wrist as much as possible, and the shoulder joint was allowed to be flexed by 160 degrees .The posture of the arm stance supported the weight using metacarpal heads, hands, and elbows, and the shoulder joints were allowed to be flexed by 90 degrees.
  Arms: Experimental group will received Comprehensive Hand Repetitive Intensive Strength Training
Other: Routine Physical Therapy — Received 60 minutes per a session, three sessions a week, at a total of 30 sessions per 10 weeks by creating a home program, which consisted of a total of 8 exercises that enhanced the muscular strength of the upper limb including the triceps brachii and extensor carpi radialis, and conveyed an effect of reaching the muscles out. flexion and extension muscle strengthening with towel, hand grip and wrist extension muscle strengthening This exercise consisted of shoulder extension muscle, elbow flexion muscle, shoulder abduction muscle, and elbow extension muscle strengthening with a thera band, as well as hand grip, forearm with a velcro board, wrist extension muscle strengthening with sandbag and shoulder abduction-extension muscle strengthening with a thera band.
  Arms: Routine Physical Therapy

SUMMARY:
Hemiplegia is the medical term for paralysis of one side of the body This means their shoulder; arm, hand, leg and foot are all completely paralyzed.. It results in muscular wasting on the affected side, impairs gait, reduces motor abilities, and causes instability and a loss of grasping capacity. The patient's quality of life is impacted by hemiplegia because it impairs brain and spinal cord functions Hemiplegic cerebral palsy is the type of cerebral palsy in which there is absolutely no use of one side of the body. This means their shoulder; arm, hand, leg and foot are all completely paralyzed. Hemiplegia in infants and children is a type of Cerebral Palsy that results from damage to the part (hemisphere) of the brain that controls muscle movements. This damage may occur before, during or shortly after birth. The term hemiplegia means that the paralysis is on one vertical half of the body.

DETAILED DESCRIPTION:
The Comprehensive Hand Repetitive Intensive Strength Training (CHRIST) program is designed to provides special training for enhancing muscular strength of the upper limb.

The current study will be a randomized control trial, and data will be collected from Ittefaq Hospital Lahore Pakistan. The study will include 30 patients equally divided into two groups experimental group included 15 patients, and the control group included 15 patients and was randomly allocated. The inclusion criteria for the study will be Comprehensive Hand Repetitive Intensive Strength Training on the upper limb of CP patients with age between 6 to 12 years and both genders will be included children who have normal communication skills and cognitive function will be included and give 30 minutes per session three sessions in a week and total 30 sessions per ten weeks and to normalize muscle tone and patient able to perform ADLS.

Children having damaged musculoskeletal system including fracture of upper limb and contracture will be excluded children having undergone administration of medicine influencing muscular strength and spasticity will be excluded tools used for data collection are Jebsen-Taylor Hand Function Test and ABIL Hand for upper limb and data will be analyzed by SPSS version 26.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6 to 12 years will be included
* Both genders will be included
* GMFCS I and II
* Children who have normal communication skills and cognitive functions will be included

Exclusion Criteria:

* Children having damage to the musculoskeletal system including fracture of the upper limb and contracture will be excluded
* Children who have undergone the administration of medicine influencing muscular strength and spasticity will be excluded

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2024-12-25 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Jebsen-Taylor Hand Function Test (JTHFT) | 15 to 30 minutes
  The Jebsen-Taylor Hand Function Test (JTHFT) is a standardized and objective measure of fine and gross motor hand function using simulated activities of daily living (ADL). The JTHFT has seven subsets which are writing, simulated page-turning, lifting small objects, stimulated tree feeding, stacking, and lifting large, lightweight, and heavy objects. [JTHFT finds easy applicability in clinical settings since it can be administered in a short time by using readily available materials. Several studies report that the JTHFT is a valid assessment tool for the measurement of hand dysfunctions from a variety of patient populations having high reliability were (0.84-0.94 )
ABIL HAND | 10 - 20 minutes
  ABILHAND-Kids Survey, which evaluates upper extremity function in children with cerebral palsy ABILHAND-Kids survey evaluates the bilateral upper extremities of children, and which has proven validity and reliability were 0.96 and 0.70 , including 21 questions for families related to the common tasks undertaken by their children in their daily living activities. The ABILHAND-Kids survey was originally developed in French as a standard means of assessment of manual ability in children with CP. This survey evaluates the most typical indicators of manual activity, in which some of the items were developed based on the ABILHAND-Kids survey, which was developed to assess manual ability in adult patients, while other items were selected from existing scales or were adapted to broaden the variability of activities

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Feroz, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kara OK, Yardimci BN, Sahin S, Orhan C, Livanelioglu A, Soylu AR. Combined Effects of Mirror Therapy and Exercises on the Upper Extremities in Children with Unilateral Cerebral Palsy: A Randomized Controlled Trial. Dev Neurorehabil. 2020 May;23(4):253-264. doi: 10.1080/17518423.2019.1662853. Epub 2019 Sep 13. PMID 31514564